CLINICAL TRIAL: NCT00005470
Title: Divergence of Blood Pressure By Race in Adolescent Girls
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4952; R01HL052911 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To continue examinations of 670 girls enrolled in the National Growth and Health Study (NGHS) for four more years, adding measurements of total peripheral resistance, cardiac output, DEXA scans for fat-free mass and fat mass, left ventricular mass and geometry, circulating blood volume, whole blood viscosity, and left ventricular contractility.

DETAILED DESCRIPTION:
BACKGROUND:

African-American women have a substantially higher prevalence of hypertension and suffer greater morbidity and mortality due to blood pressure elevation than white-American women. Much of this ethnic difference in blood pressure is due to increased obesity in African-American women. In contrast, young African-American and white-American girls have similar levels of obesity and blood pressure. The hemodynamic changes that occur with developing obesity and result in this ethnic difference in blood pressure have not been well characterized. Cross-sectional studies of adolescents have shown that despite similar blood pressure levels, African-Americans have higher total peripheral resistance while whites have higher cardiac output. Cross-sectional studies of adults show that obesity is associated with elevation of cardiac output. If such an obesity-related increase in cardiac output is superimposed on the underlying elevation of total peripheral resistance in African-American girls, these hemodynamic factors could be responsible for the developing ethnic divergence in blood pressure seen in late adolescence as African-American girls develop an increasing prevalence and severity of obesity.

This investigation will provide important new knowledge regarding the longitudinal changes and interrelationships among the potential hemodynamic factors which define the association between developing obesity and blood pressure elevation. In the clinical setting where obesity is very difficult to prevent or treat, it is important to understand the mechanisms by which obesity results in elevated blood pressure. The results of this cohort study will provide the basis for rational and specific clinical strategies to interrupt the pathophysiologic process by which obesity leads to hypertension and places African-American women at particularly increased risk for cardiovascular disease morbidity and mortality.

The NGHS was initiated by the NHLBI in 1985 as a contract-supported program to determine if the Black-white differences in the development of obesity in 2,379 pubescent females were due to differences in psychosocial, socioeconomic and other environmental factors. The study also sought to determine whether differences in the development of obesity led to Black-white differences in other coronary heart disease risk factors, such as blood pressure and serum lipids. The study has been renewed twice, the last time as an investigator-initiated study. See the National Growth and Health Study for the complete write-up.

DESIGN NARRATIVE:

The ancillary study is a prospective cohort study of 355 African-American and 315 white-American females from the NHLBl Growth and Health Study as these women progress from age 18-19 years to age 21-22 years. The study includes yearly measurement of anthropometrics, blood pressure, and echocardiographic determination of cardiac output and total peripheral resistance. In addition, factors which may relate to changes in cardiac output and total peripheral resistance, such as circulating blood volume (left ventricular end-diastolic volume), heart rate, left ventricular contractility, whole blood viscosity, and left ventricular mass and geometry are measured.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Daniels — Children's Hospital & Medical Center

REFERENCES:
- [Background] Kimm SY, Glynn NW, Aston CE, Poehlman ET, Daniels SR. Effects of race, cigarette smoking, and use of contraceptive medications on resting energy expenditure in young women. Am J Epidemiol. 2001 Oct 15;154(8):718-24. doi: 10.1093/aje/154.8.718. PMID 11590084